CLINICAL TRIAL: NCT00000694
Title: A Phase I Trial of Recombinant Human Granulocyte-Macrophage Colony Stimulating Factor (rHuGM-CSF), Recombinant Alpha Interferon and Azidothymidine (AZT) in AIDS-Associated Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 090; 11065 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Interferon Alfa-2b; Immune System; Drug Evaluation; Drug Therapy, Combination; Granulocyte-Macrophage Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Interferon alpha-2; Zidovudine; sargramostim

INTERVENTIONS:
Drug: Interferon alfa-2b
Drug: Zidovudine
Drug: Sargramostim

SUMMARY:
To define the best doses of sargramostim ( granulocyte-macrophage colony-stimulating factor; GM-CSF ), interferon alfa-2b ( IFN-A2b ), and zidovudine ( AZT ) to give together in patients with AIDS-associated Kaposi's sarcoma ( KS ), to learn about the side effects of these drugs when they are given together for 8 weeks, and to find out whether the combination of GM-CSF, IFN-A2b, and AZT has any effect on KS, HIV, or the immune system.

Studies show that IFN-A2b can cause KS tumors to shrink or disappear in about 30 percent of patients. IFN-A2b can greatly reduce the growth of the HIV virus in test tube experiments and perhaps in patients. AZT has also been shown to reduce the growth of HIV and show improvements in the immune system with fewer infections. Test tube experiments show that when IFN-A2b and AZT are used together, they reduce the growth of the HIV virus much more effectively than when either drug is used alone. In recent studies of the combination of interferon alpha and AZT in patients with KS, more than 40 percent of the patients showed shrinkage of their tumors, and some showed evidence for suppression of HIV growth in the body. However, the combination of IFN-A2b with AZT often caused a marked lowering of the white blood cell (WBC) count, especially a type of WBC called the granulocyte (or neutrophil) which is important in the body's defense against infection. Recombinant human GM-CSF is a human protein which is produced in bacteria. It has been shown to cause an increase in the WBC count.

DETAILED DESCRIPTION:
Studies show that IFN-A2b can cause KS tumors to shrink or disappear in about 30 percent of patients. IFN-A2b can greatly reduce the growth of the HIV virus in test tube experiments and perhaps in patients. AZT has also been shown to reduce the growth of HIV and show improvements in the immune system with fewer infections. Test tube experiments show that when IFN-A2b and AZT are used together, they reduce the growth of the HIV virus much more effectively than when either drug is used alone. In recent studies of the combination of interferon alpha and AZT in patients with KS, more than 40 percent of the patients showed shrinkage of their tumors, and some showed evidence for suppression of HIV growth in the body. However, the combination of IFN-A2b with AZT often caused a marked lowering of the white blood cell (WBC) count, especially a type of WBC called the granulocyte (or neutrophil) which is important in the body's defense against infection. Recombinant human GM-CSF is a human protein which is produced in bacteria. It has been shown to cause an increase in the WBC count.

AMENDED: 900910 to allow one patient to be treated beyond one year. Original design: GM-CSF, IFN-A2b, and AZT are given every day for 8 weeks. There are 6 patients per dose level. IFN-A2b and GM-CSF are given in two separate injections under the skin (subcutaneous injection) once a day. AZT is given orally every 4 hours (6 times/day). The first patients are given doses of the drugs that are quite well tolerated when given alone. If these dosages are tolerated without serious side effects, the dosage of IFN-A2b is increased in subsequent groups of patients. Maintenance treatment consisting of the same dose received at the conclusion of the initial 8 week course of treatment will be resumed with eligible patients for up to 1 year.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis for Pneumocystis carinii pneumonia (PCP) with aerosolized pentamidine. Ibuprofen, not to exceed 1600 mg/day, for fever or analgesia.

Biopsy-proven Kaposi's sarcoma confined to the skin, lymph nodes, or non-nodular lesions of the hard palate. Positive antibody to HIV confirmed by any federally licensed ELISA test kit. Patients must be able to give informed consent.

* Allowed: Basal cell carcinoma.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Prior or concurrent opportunistic infection or B symptoms (unexplained fever, night sweats, > 10 percent involuntary weight loss or diarrhea persisting > 2 weeks).
* Visceral (non-nodal) Kaposi's sarcoma including extensive oral lesions.
* Severe (> 2+) tumor-associated edema.
* Concurrent neoplasia (excluding basal cell carcinoma).
* Significant cardiac disease (New York Heart Association class III or IV) or history of myocardial infarction o significant cardiac arrhythmias.
* Dementia (= or > stage 2).

Concurrent Medication:

Excluded:

* Any systemic chemoprophylaxis not specifically allowed.
* Aspirin and acetaminophen.
* Nonsteroidal anti-inflammatory agents not specifically allowed.
* Corticosteroids.
* Barbiturates.
* Other antiviral agents, immunotherapy, hormonal therapy, chemotherapy directed at treatment of viral infection or malignancy.
* Other investigational agents.

Concurrent Treatment:

Excluded:

* Radiation therapy directed at treatment of viral infection or malignancy.

Patients with the following are excluded:

* Prior or concurrent opportunistic infection or B symptoms (unexplained fever, night sweats, > 10 percent involuntary weight loss or diarrhea persisting > 2 weeks).
* Visceral (non-nodal) Kaposi's sarcoma including extensive oral lesions.
* Severe (> 2+) tumor-associated edema.
* Concurrent neoplasia (excluding basal cell carcinoma).
* Significant cardiac disease (New York Heart Association class III or IV) or history of myocardial infarction or significant cardiac arrhythmias.
* Dementia (= or > stage 2).

Prior Medication:

Excluded:

* Interferon alpha-2b.
* Granulocyte-macrophage colony-stimulating factor (GM-CSF).
* Prior grade 3 or grade 4 toxicity during AZT therapy.
* Excluded within 30 days of study entry:
* Zidovudine (AZT).
* Corticosteroids.
* Biologic response modifiers.
* Cytotoxic chemotherapy.
* Antiretroviral agents.
* Toxicity grades according to NIAID Recommendations for Grading Acute and Subacute Toxic Effects (Adults).

Prior Treatment:

Excluded within 30 days of study entry:

* Requirement for red blood cell transfusions within 30 days of study entry.
* Radiation therapy.

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Study Completion 1992-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SE Krown, Study Chair
Locations (1):
- Mem Sloan - Kettering Cancer Ctr, New York, New York, United States

REFERENCES:
- [Background] Krown SE, Paredes J, Bundow D, Polsky B, Gold JW, Flomenberg N. Interferon-alpha, zidovudine, and granulocyte-macrophage colony-stimulating factor: a phase I AIDS Clinical Trials Group study in patients with Kaposi's sarcoma associated with AIDS. J Clin Oncol. 1992 Aug;10(8):1344-51. doi: 10.1200/JCO.1992.10.8.1344. PMID 1634925
- [Background] Krown SE, Paredes J, Bundow D, Flomenberg N. Combination therapy with interferon-alpha (IFN-alpha), zidovudine (AZT), and recombinant granulocyte-macrophage colony-stimulating factor (GM-CSF): a phase I trial in patients with AIDS-associated Kaposi's sarcoma. Int Conf AIDS. 1990 Jun 20-23;6(3):214 (abstract no SB513)